CLINICAL TRIAL: NCT06304337
Title: Randomized Controlled Clinical Study of the Incidence of Hypoxia in a Novel Oropharyngeal Airway During Painless Gastroenteroscopy
Brief Title: Application of New Oropharyngeal Airway Management in Patients Undergoing Painless Gastroenteroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YXLL-KY-2023(162)
Record Dates: First submitted 2024-01-29; First posted 2024-03-12 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Airway Management

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ordinary oral cushion set (No Intervention): Before anesthesia induction, patients in the experimental group received 5-6L/min of oxygen for about 1min through the endoscopic bite connecting oxygen supply device, and patients in the control group inhaled 5-6L/min of oxygen for about 1min through the nasal catheter.Both groups were anesthetised with propofol 3mg/Kg and sufentanil 7ug.Sufentanil was given at the beginning of pre-oxygen inhalation, and propofol was given 1min later. After the subjects achieved sufficient sedation (about BIS40), The ordinary endoscopic bite group began to perform endoscopic operation after sufficient sedation was achieved,In both groups, 5mg/Kg/h propofol was continuously pumped to maintain anesthesia until completion of the examination.
- New oropharyngeal airway group (Experimental): Before anesthesia induction, patients in the experimental group received 5-6L/min of oxygen for about 1min through the endoscopic bite connecting oxygen supply device, and patients in the control group inhaled 5-6L/min of oxygen for about 1min through the nasal catheter.Both groups were anesthetised with propofol 3mg/Kg and sufentanil 7ug.Sufentanil was given at the beginning of pre-oxygen inhalation, and propofol was given 1min later. After the subjects achieved sufficient sedation (about BIS40), the new oropharyngeal airway group was placed into the oropharyngeal airway through the endoscopic bite and then began gastroscopy,In both groups, 5mg/Kg/h propofol was continuously pumped to maintain anesthesia until completion of the examination
  Interventions: Device: New oropharyngeal airway group

INTERVENTIONS:
Device: New oropharyngeal airway group — Oropharyngeal airwayIt is composed of nasal plug, bite mouth, oropharyngeal passage, oxygen supply tube, rope and optional accessories carbon dioxide gas catheter and carbon dioxide collection tube.For patients undergoing endoscopic surgery/examination to prevent airway obstruction caused by backtongue fall, establish oropharyngeal airway for patients, and provide nasal oxygen at the same time, JK model can monitor oropharyngeal end-expiratory carbon dioxide collection.
  Arms: New oropharyngeal airway group

SUMMARY:
The objective of this study was to investigate the application of new oropharyngeal airway management in patients undergoing painless gastroenteroscopy.To see if it can really solve the problem of airway obstruction during anesthesia.The incidence of hypoxia (Spo2<90%, t>10s) and severe hypoxia (Spo2<85%) during anesthesia and sedation, as well as the incidence of cough and laryngeal spasm, as well as the dose, endoscopist satisfaction, and the incidence of various adverse events were observed.To accumulate clinical experience and reference of anesthesia in obese patients.

DETAILED DESCRIPTION:
Painless endoscopy is a popular method of endoscopic diagnosis and treatment.General intravenous anesthesia with propofol and fentanyl has been widely used in painless endoscopic diagnosis and treatment.However, the combined application of the two has an obvious respiratory central inhibitory effect, resulting in a decrease in blood oxygen saturation in patients, especially in obese and elderly patients, who are more prone to a sudden decrease in blood oxygen, and even life-threatening.Due to the potential risk of upper airway obstruction in some obese patients, intraoperative hypopnea may occur during painless colonoscopy due to sedative and analgesic drugs.Causing the patient to be starved of oxygen.At present, there is no special oropharyngeal ventilation device for gastroenteroscopy.In recent years, a new type of oropharyngeal ventilation channel has been developed and applied in clinic.Compared with the traditional nasal catheter, the new oropharyngeal airway nasal mask can better fit the patient's face, ensure the internal air tightness of the nose mask, and maximize the oxygen supply efficiency.Connecting the carbon dioxide outlet of the oral pharyngeal airway body can not only collect the exhaled gas of the patient, but also reduce the backflow of carbon dioxide gas.It can also be connected to a carbon dioxide detection device to monitor the partial pressure of carbon dioxide at the end of a patient's breath in real time.To evaluate whether a new type of oropharyngeal airway can reduce the incidence of hypoxia during painless gastroenteroscopy in general patients, the investigators present this study and investigate the safety and efficacy of the new type of oropharyngeal airway.

ELIGIBILITY:
Inclusion Criteria:Voluntary acceptance;Asa1-2 level;Age 18-95y;Mallampati grades Ⅰ or Ⅱ

Exclusion Criteria:

1. Patients with blood clotting disorders or a tendency to oropharyngeal bleeding, mucosal damage or space occupation, difficulty in placing oropharyngeal airway, etc., who cannot perform oropharyngeal airway ventilation;
2. Severe cardiac insufficiency (<4mets);
3. Patients with severe renal insufficiency (requiring dialysis before surgery);
4. Diagnosed severe liver insufficiency;
5. Diagnosed with chronic obstructive pulmonary disease (COPD) or currently suffering from other acute or chronic lung diseases, requiring long-term or intermittent oxygen therapy;
6. Increased intracranial pressure;
7. Upper respiratory tract infections such as mouth, nose or throat;
8. Fever (core body temperature >37.5 degrees Celsius);
9. a confirmed diagnosis of pregnancy or breastfeeding;
10. Allergic to sedatives such as propofol or equipment such as tape;
11. Emergency surgery;
12. Multiple trauma;
13. SpO2 < 95% in preoperative breathing air;

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2025-03-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxia (Spo2<90%,t>10s) and severe hypoxia (Spo2<85%) during anesthetic sedation | during surgery
  The incidence of hypoxia (75%≤SpO2 < 90%, < 60s) and severe hypoxia (SpO2 < 75% or 75%≤SpO2 < 90%, ≥60s) during anesthesia was recorded,The time of intervention was half or disappearance of end-expiratory carbon dioxide and/or disappearance of thoracic fluctuation and/or SpO2 < 95%, that is, open airway manipulation was taken successively until SpO2≥95%, and the last means of opening the airway was recorded.The means of opening the airway of the two groups were the same, including: 1) adjusting the oxygen flow;2) Lift the lower jaw;3) Mask ventilation (pull out the gastroscope if necessary);4) Tracheal intubation or laryngeal mask for ventilator assisted ventilation.

SECONDARY OUTCOMES:
The incidence of choking, reflux aspiration and laryngeal spasm were recorded | during surgery
  The incidence of choking, reflux aspiration and laryngeal spasm were recorded
The dose of additional drugs during the operation | during surgery
  The total amount of propofol administered throughout the test was recorded
Endoscopist satisfaction | within 30 minutes after surgery
  The endoscopist was asked to score the satisfaction after the operation
Record adverse events that occur throughout the process | during surgery
  Apnea or slow breathing episodes (defined as respiratory rate <6 beats/min);Bradycardia is defined as a heart rate <50 beats/min.Serious adverse events such as tracheal intubation, non-invasive ventilation, use of vasopressors, and hospitalization are required.

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Wu, Study Director — Department director
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University（Qianfoshan Hospital, Shandong Province）, Jinan, China

IPD SHARING:
Plan to Share IPD: No